CLINICAL TRIAL: NCT05375864
Title: Prognostic Impact of Early Oseltamivir Carboxylate Low Plasma Concentration in Critically Ill Patients With Severe Influenza: a Prospective Cohort Study
Brief Title: Early Oseltamivir Carboxylate Low Plasma Concentration in Patients Admitted to Intensive Care for Severe Influenza
Acronym: OPTIFLU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP210090; 2022-002377-28 (EudraCT Number)
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Severe Influenza
Keywords: Influenza; Intensive Care Unit; oseltamivir; paracetamol absorption test
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Masking Description: 1. Laboratory staff assessing the paracetamol assay will be blinded to the results of the plasma oseltamivir assay and vice versa.
  2. The investigators will be blinded to the assays.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paracetamol absorption test (Experimental)
  Interventions: Other: Absorption test

INTERVENTIONS:
Other: Absorption test — Paracetamol's administration (1 gram) - 48 hours after oseltamivir administration.

SUMMARY:
Introduction

Pandemic and seasonal influenza epidemics can be associated with a high degree of morbidity and mortality, especially in patients developing severe influenza pneumonitis with the acute respiratory distress syndrome (ARDS) or the less frequent fulminant myocarditis. Early administration (i.e. in the first 48 hours) of the neuraminidase inhibitor oseltamivir is associated with reduced mortality in patients hospitalized for severe influenza. Early oseltamivir administration, which can only be given orally (or through a nasogastric tube), is thus recommended by the World Health Organization in patients hospitalized for severe influenza, including those requiring intensive care (ICU) admission. However, enteric absorption may be compromised in critically ill patients due to impaired gut function.

Hypothesis/Objective

The hypothese is that, in patients admitted for severe influenza, early (i.e., measured at the 48th hour of treatment initiation) oseltamivir carboxylate (OC) low plasma concentration would be: 1) associated with a poor prognosis; and 2) detectable by carrying out a paracetamol absorption test (PAT).

The main objective of the study is to determine the prognostic impact of early OC low plasma concentration in patients admitted to the intensive care unit (ICU) for severe influenza.

Primary outcome measure: Number of live ventilator-free days at 28-day in patients with versus without OC low plasma concentration.

DETAILED DESCRIPTION:
Methods

Prospective cohort study conducted in 22 French intensive care units. Adult patients admitted to the ICU for severe influenza requiring invasive mechanical ventilation and treated with oseltamivir through a gastric tube for less than 24 hours will be included.

After inclusion, oseltamivir treatment will be continued through a gastric tube (75mg x 2 /day). After the 4th administration, plasma peak concentration of oseltamivir phosphate (OP) will be dosed at 60 minutes (CmaxOP) and plasma residual concentration of OC will be dosed at 12 hours (just before the 5th dose) (CresOC). A paracetamol absorption test will also be performed at the same time (consisting in the measurement of plasma paracetamol concentration 60 minutes after enteral loading with 1000 mg of paracetamol). CmaxOP and CresOC will also be measured at day 3 and 5 in order to realize pharmacokinetic analysis. Nasal swabs will be performed at inclusion (day 1) and day 5 for viral load quantification and viral strain sequencing (detection of the H275Y mutation). Clinical and biological variables will be collected from day 1 to day 90.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Confirmed severe influenza infection requiring intensive care with tracheal intubation for invasive mechanical ventilation (influenza ARDS with or without bacterial co-infection, cardiorespiratory decompensation of influenza origin, influenza myocarditis)
* Oseltamivir treatment administered through a gastric tube initiated since less than 24 hours (i.e. maximum two doses administered)
* Affiliation to a social security system or beneficiary (excluding AME)
* Written consent obtained (or under emergency procedures)

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Weight less than 40 kg
* Zanamivir or other antiviral effective treatment received for more than 24 hours
* Other respiratory virus infection (including SARS-CoV-2)
* Contra-indication to esophageal tube insertion or use
* Child-Pugh C cirrhosis or severe liver insufficiency
* Paracetamol allergy
* Ongoing participation in an interventional therapeutic trial (medicine that may interact with paracetamol or oseltamivir)
* Patient benefiting from AME (State Medical Aid)
* Patient deprived of liberty or under legal protection (guardianship or curatorship)
* For patients not included in an emergency situation: Inability, according to the investigator, to understand or refusal to sign the informed consent to participate in the study (non-French-speaking patient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Live ventilator-free days (VFDs) | Day 28
  VFDs = 0 if subject dies within 28 days of mechanical ventilation. VFDs = 28 - x if successfully liberated from ventilation x days after initiation.
  VFDs = 0 if the subject is mechanically ventilated for > 28 days.

SECONDARY OUTCOMES:
Diagnostic performance of the paracetamol absorption test (PAT) | 48 hours
  Sensitivity = ability of PAT to correctly classify a patient as "having a low oseltamivir carboxylate (OC) concentration" = (true positive) / (true positive + false negative) Specificity = ability of PAT to correctly classify a patient as "not having a low oseltamivir carboxylate (OC) concentration" = (true negative) / (true negative + false positive) Positive predictive value (PPV) = percentage of patients with negative PAT who actually are "having a low oseltamivir carboxylate (OC) concentration"= (true positive) / (true positive + false positive) Negative predictive value (NPV) = percentage of patients with positive PAT who actually are not ""having a low oseltamivir carboxylate (OC) concentration" = (true negative) / (false negative + true negative) Positive Likelihood Ratio = Sensitivity / (1 - Specificity) Negative Likelihood Ratio = (1 - Sensitivity) / Specificity
Prevalence of patients with low plasma OC concentration | 48 hours
Independent variables present on admission associated with low plasma OC concentration | 48 hours
Prevalence of acquisition early OC concentration and viral clearance | 48 hours
Prevalence of acquisition of the oseltamivir resistance mutation (H275Y) in patients with versus without low plasma OC concentration. | 48 hours and day 5
Maximum oseltamivir carboxylate concentrations measurement | Days 2, 3 and 5
Maximum oseltamivir phosphate concentrations measurement | Days 2, 3 and 5
Residual oseltamivir carboxylate concentrations measurement | Days 2, 3 and 5
Residual oseltamivir phosphate concentrations measurement | Days 2, 3 and 5
Mortality | Days 28 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Fleur Haudebourg, M.D, Study Director — Assistance Publique Hôpitaux de Paris - CHU Henri Mondor
Locations (1):
- Anne-Fleur Haudebourg, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWNED BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION